CLINICAL TRIAL: NCT02593695
Title: Deep Brain Stimulation of Nucleus Accumbens as a New Treatment to Treat Severe Anorexia Nervosa
Brief Title: Deep Brain Stimulation of Nucleus Accumbens to Treat Severe Anorexia Nervosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Guodong Gao, Neurosurgery Department, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANDBS
Record Dates: First submitted 2015-10-14; First posted 2015-11-02 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Deep Brain Stimulation; Nucleus accumbens
MeSH Terms: conditions — Anorexia Nervosa | interventions — Deep Brain Stimulation; Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Continuous deep brain stimulation of bilateral nucleus accumbens
  Interventions: Procedure: Deep brain stimulation
- Standard Control (Active Comparator): Fluoxetine
  Interventions: Other: Fluoxetine

INTERVENTIONS:
Procedure: Deep brain stimulation — Deep brain stimulation of bilateral nucleus accumbens
  Other Names: DBS
  Arms: Deep Brain Stimulation
Other: Fluoxetine — Fluoxetine is one of selective serotonin reuptake inhibitors(SSRIs).
  Arms: Standard Control

SUMMARY:
Anorexia nervosa (AN) is a complex and severe psychiatric disorder with high relapse rates under standard treatment.Deep brain stimulation (DBS) may be a novel treatment in severe Anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years of age, male or female patients.
2. Diagnosis is Anorexia Nervosa(AN) by the DSMIV(Diagnostic and Statistical Manual of Mental Disorders Fourth Edition).
3. BMI<16.
4. Long-term pharmacotherapy resistance.
5. Written informed consent.
6. normal intelligence and compliance

Exclusion Criteria:

1. Surgical contradiction（implanted artificial cochlea、cardiac pacemaker、cardiac defibrillator、stereotactic ablative surgery、DBS）or receive other surgery which may influence this time of surgery in half year, or other neurosurgical contradictions； History of brain trauma；
2. History of severe neuropsychiatric disease；
3. Epilepsy；
4. severe liver、kidney、heart and lung disease, severe hypertension and severe orthostatic hypotension；
5. Severe diabetes ,severe cardiovascular and cerebrovascular disease；
6. Malignant tumor；
7. Being using anticoagulant or showing clinical hemorrhagic tendency； Pregnant female；
8. Patients are taking part in other clinical trials in recent 3months； Being deem as unfit for the trials by researcher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
BMI | 6 month

SECONDARY OUTCOMES:
weight | 6 month
Yale-Brown Obsessive Compulsive Scale | 6 month
  Yale-Brown Obsessive Compulsive Scale(Y-BOCS) is used to evaluate obsessive compulsive symptom.
Self-Rating Depression Scale | 6 month
  Self-Rating Depression Scale(SDS) is used to evaluate depression symptom.
The Symptom Checklist-90 | 6 month
  The Symptom Checklist-90(SCL-90) is used to evaluate general status.

CONTACTS AND LOCATIONS:
Overall Officials: Guo-dong Gao, M.D., Principal Investigator — Department of neurosurgery, Tangdu Hospital
Locations (1):
- Department of neurosurgery, Tangdu Hospital, Xi'an, Shaanxi, China